| Perfusionsindex som ma | arkør for nerfusion | og flow ved indledning a | f anæstesi v1.0 05032019 |
|---|---|---|---|

# **Protokol**

# Perfusionsindex som markør for perfusion og flow ved indledning af anæstesi

Version 1.0

05032019

Ovl. Jakob Højlund, Anæstesiologisk afdeling, Hvidovre Hospital

AutorisationsID 00V8C

| Perfusionsindex som markør for perfusion | n og flow ved | ed indledning at | t anæstesi vl.0 | 05032019 |
|---|---|---|---|---|
|---|---|---|---|---|

### **Protokol**

# Perfusionsindex som markør for perfusion og flow ved indledning af anæstesi

Ansvarlig læge: Ovl. Jakob Højlund, Anæstesiologisk afdeling, Hvidovre Hospital

# Baggrund og formål:

Perioperativ hæmodynamisk monitorering har traditionelt betjent sig af simple og for-hånden-værende parametre som blodtryk og hjertefrekvens. Nyere tilgange tilstræber en indgangsvinkel som er mere orienteret mod (optimering af) systemisk blood flow (Vincent et al. Critical Care (2015) 19:224). Det reelle fokus burde dog ideelt være på perfusionen af organerne, men dette har ikke vundet synderligt indpas, idet der ikke har eksistereret enkle og billige metoder til dette (Dyson and Singer, Curr Opin Crit Care (2011) 17:281). Perfusionsindex (PI) kan opnås simpelt og non-invasivt vha. puls-oximetri, som allerede er standard monitorering i det perioperative forløb. Perfusionsindex opnås via fotopletysmografi/pulsoxymetri og er et simpelt forholdstal som angiver hvor stor en del af signalet (reelt: signalsvækkelsen) der er pulsatilt. Perfusionsindexet er en prædiktor for komplikationsfrekvensen ved større kirurgi (van Genderen et al. Crit Care. 2014; 18(3): R114) samt mortaliteten hos akut indlagte kritisk syge patienter (Oskay et al. Am J Emerg Med. 2015 Aug;33(8):1042-4). Samtidigt er ændringer i perfusionsindex en tidlig prædiktor for hypovolæmi hos raske forsøgspersoner (van Genderen et al. Anesth Analg (2013) 116:351–6). Der findes ikke litteratur angående perfusionsindexet ifm indledning af anæstesi.

Et anæstesiforløb i fuld bedøvelse kan være præget af negativ påvirkning af kredsløbet. Specielt indledningsfasen kan være kritisk. Standard-monitorering består af intermitterende blodtryksmåling, hvorfor en kontinuert overvågning kunne være ønskværdig. De gængse metoder til dette er desværre dyre eller noget besværlige at anvende rutinemæssigt. Vi håber at måling af Perfusionsindexet kan give en tidlig advarsel om kredsløbet er ustabilt og således medvirke til en endnu bedre og sikrere behandling af patienter der skal i fuld bedøvelse.

Hypotese, endpoints, rationale: Monitorering af perfusionsindex kan give værdifuld information om den systemiske hæmodynamik under indledningen af generel anæstesi. Forsøget vil søge at redegøre for sammenhænge mellem ændringer i hjertets slagvolumen, blodtryk og perfusionsindex under indledningen

#### Perfusionsindex som markør for perfusion og flow ved indledning af anæstesi\_v1.0\_05032019

af generel anæstesi. Studiet er eksplorativt, altså uden veldefinerede outcome mål. Vi forventer dog specielt fokus på udgangsværdier: "høj" vs "lav" samt trends ifm anæstesiindledningen: "bevaret eller stigende" vs "faldende". Kan metoden valideres kan dette potentielt komme et stort antal patienter til gode idet mere avancerede metoder er invasive, besværlige og omkostningstunge og således forbeholdt et fåtal af "højrisiko" patienter.

## Metodologi:

Design: Observationelt kvalitetssikrings projekt.

Sted for undersøgelsen: Operationsgangen, COP, Hvidovre Hospital

Metode: Deskriptivt studie. 40 patienter.

Tidsperiode: Inklusion og dataindsamling forventes at foregå fra 1. maj 2019 til 30. juni 2020.

Procedure: Alle patienter som skal i generel anæstesi monitoreres rutinemæssig med pulsoxymetri, EKG samt non-invasivt intermitterende blodtryk. I forbindelse med studiet vil patienterne tillige blive monitoreret med endnu et pulsoxymeter (Masimo Radical 7) samt LiDCO CNAP monitor. Begge apparater er CE-godkendt. Det drejer som en en ikke stram klemme som sidder på en finger, respektivt to små blodtryksmanchetter som sidder på to andre fingre. Dette vil intet ubehag og ingen risiko medføre. Patienternes behandling vil være som vanligt og projektet medfører ingen ekstra interventioner for patienterne. Der vil ikke blive udtaget biologisk materiale i forbindelse med undersøgelsen. De inkluderede patienter ikke blive udsat for intervention ud over vanlig klinisk praksis og behandling på afdelingen.

Statistik: Idet forsøget er et deskriptivt kohortestudie med en nyere monitoreringsmodalitet kendes hverken forventet spredning eller varians for data. Det er således ikke muligt at udføre en styrkebergning. Vi ønsker at inkludere 40 patienter.

Analyse: Ud fra præliminære observationer forventer vi at stratificere patienterne efter "højt" resp. "lavt" perfusionsindex før anæstesi-indledningen. For disse grupper vil vi undersøge den prædiktive værdi af "bevaret/stigende" vs. "faldende" perfusionsindex efter anæstesiindledning til at forudse ustabilt kredsløb.

Patientpopulation: Patienter som er planlagt til operation i generel anæstesi (fuld bedøvelse).

Inklusionskriterier: Patienter som undergår planlagt kirurgi under generel anæstesi. Patienterne vil blive informeret om undersøgelsen og skal give informeret samtykke for at blive inkluderet.

Eksklusionskriterier: Børn. Gravide. Inhabile.

Risici, bivirkninger og ulemper: Som beskrevet medfører den ekstra monitorering hverken ulemper, risici eller bivirkninger for de inkluderede patienter.

Etiske aspekter: Idet forsøget indebærer yderligere, men risikofri, monitorering, vil forsøgsdeltagerne ingen risiko løbe ved deltagelse. Vi håber at resultaterne vil komme fremtidige patienter til gode.

#### Perfusionsindex som markør for perfusion og flow ved indledning af anæstesi\_v1.0\_05032019

Dataregistrering: Patienterne identificeres ved hjælp af et tildelt unikt forsøgsspecifikt id-nummer. Efter informeret samtykke opsamles fra journalen udelukkende følgende baggrundsdata: Alder, højde, vægt, køn, samt basal nosografisk information i punktform (fx hypertension, velbehandlet; diabetes type 2, o.s.v.). Dette fremgår af deltagerinformationen. Ved undersøgelsens afslutning bliver alle personidentificérbare data destrueret. Oplysningerne om forsøgspersonerne behandles efter lov om behandling af personoplysninger. Forsøget er anmeldt til Datatilsynet under Region Hovedstadens paraplyanmeldelse: AHH-20146-094.

Initiativ til forsøget kommer fra den forsøgsansvarlige læge. Forsøget vil udelukkende blive finansieret af Anæstesiologisk afdeling, Hvidovre Hospital.

Der vil ikke blive udbetalt vederlag til patienterne.

Procedurer for skriftlig og mundtlig information samt informeret samtykke: Skriftlig deltagerinformation vil blive udleveret hurtigst muligt efter at patienten identificeres som opfyldende inklusionskriterierne, typisk i forbindelse med at deltagerne bookes til operation; ellers snarest herefter. Mundtlig information og samtykke til inklusion vil foregå senere ved det præanæstesiologiske tilsyn forud for operationen. Denne samtale foregår uforstyrret i aflukket lokale. Skulle patienten ønske det er der mulighed for bisidder ved denne samtale. Samtykke vil søges indhentet i forbindelse med den mundtlige information. Såfremt deltageren skulle have behov for længere betænkningstid er dette muligt. Samtykke vil så blive indhentet på individualiseret tidspunkt; senest om morgenen på operationsdagen. Samtykket kan på ethvert tidspunkt trækkes tilbage.

Typisk vil der være mindst et døgns betænkningstid; men idet deltagelse er både risiko- og smertefri, finder forsøgsansvarlige det etisk acceptabelt at afvige fra dette hvis omstændighederne tilsiger dette.

Publikation: Såvel positive, negative som inkonklusive resulater vil blive søgt publiceret i relevant peerreviewed tidsskrift. Forsøget vil endvidere blive registreret og dokumenteret i clinicaltrials.gov

Videnskabsetik: Forsøget er ufarligt for deltagerne og resultaterne kan på sigt vise sig brugbare i forbindelse med de fleste generelle anæstesier i DK (ca. 400.000/år). Etisk findes forsøget aldeles berettiget.

Patienterne vil være omfattet af patienterstatningen uanset deres deltagelse i dette forsøg.